CLINICAL TRIAL: NCT03733652
Title: Study on the Optimal Treatment for Poor Efficacy of Entecavir in Chronic Hepatitis B Patients
Brief Title: Optimal Treatment for Poor Efficacy of Entecavir in Chronic Hepatitis B Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liang Peng, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PL3
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Chronic Hepatitis b; Efficacy, Self
Keywords: Chronic Hepatitis B; entecavir
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Interferon alpha-2; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tenofovir (No Intervention): Patents are treated with oral tenofovir 300mg once per day for 48 weeks. Then, tenofovir will be stopped if there is HBsAg clearance. Else, oral tenofovir 300mg once per day will be continued if HBsAg is positive.
- Interferon alfa (Active Comparator): Patents are treated with interferon alfa 2a 180μg hypodermic injection once per week for 48 weeks. Then, interferon alfa 2a will be stopped if there is HBsAg clearance. Else, oral tenofovir 300mg once per day will be used if HBsAg is positive.
  Interventions: Drug: Interferon Alfa 2a

INTERVENTIONS:
Drug: Interferon Alfa 2a — Patents are treated with interferon alfa 2a 180μg hypodermic injection once per week for 48 weeks. Then, interferon alfa 2a will be stopped if there is HBsAg clearance. Else, oral tenofovir 300mg once per day will be used if HBsAg is positive.
  Other Names: Pegasys
  Arms: Interferon alfa

SUMMARY:
There are chronic hepatitis B patients with poor antiviral efficacy of entecavir in clinical practice. Tenofovir or interferon alfa is the optimal choice right now. The aim of this study is to investigate the therapeutic effect of using tenofovir of interferon alfa in these patients.

DETAILED DESCRIPTION:
There are chronic hepatitis B patients with poor antiviral efficacy of entecavir in clinical practice. Poor efficacy is defined as hepatitis b virus DNA is still positive and decreases > 2 lg from baseline. Sequential therapy by using tenofovir or interferon alfa is the optimal choice right now. 100 patients with poor antiviral efficacy of entecavir will be recruited in this study. They are randomly divided into tenofovir group or interferon alfa group. The aim of this study is to investigate the therapeutic effect of using tenofovir of interferon alfa in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Hepatitis b virus DNA or HBsAg positive for over half a year;
2. Age from 18 to 65;
3. With poor efficacy of entecavir: Hepatitis b virus DNA is still positive at 24 weeks, and decrease > 2 lg from baseline .
4. Not be treated with interferon alfa ever before.

Exclusion Criteria:

1. Other active liver diseases;
2. Cirrhosis, hepatocellular carcinoma or other malignancy;
3. Pregnancy or lactation;
4. Human immunodeficiency virus infection or congenital immune deficiency diseases;
5. Severe diabetes, autoimmune diseases;
6. Other important organ dysfunctions;
7. Patients can not follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-15 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
HBsAg decrease after 48 weeks treatment | 48 weeks
  The patients recruited will be treated with tenofovir or interferon alfa. After 48 weeks treatment, level of HBsAg will be tested again. The investigators want to know the rate of patients with HBsAg level that decreases more than 2 lg from baseline.

SECONDARY OUTCOMES:
HBsAg clearance after 48 weeks treatment | 48 weeks
  The patients recruited would be treated with tenofovir or interferon alfa. After 48 weeks treatment, level of HBsAg will be tested again. The investigators want to know the rate of patients with HBsAg clearance which is lower than 0.05 IU/ml.
Undetectable hepatitis b virus DNA after 48 weeks treatment | 48 weeks
  The patients recruited would be treated with tenofovir or interferon alfa. After 48 weeks treatment, level of hepatitis b virus DNA will be tested again. The investigators want to know the rate of patients with undetectable hepatitis b virus DNA which is lower than 20 IU/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Peng, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided